CLINICAL TRIAL: NCT07371962
Title: "Everyone is a Hope Builder" Project Study- Therapeutic Song-writing Program
Brief Title: Sound Bite-- a Therapeutic Song-writing Program
Acronym: Sound Bite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: The Salvation Army, Hong Kong and Macau Command (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-STA-00001726
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depression
Keywords: Young people; Depression; Therapeutic song-writing; Self-stigma; Hope; Randomized Control Trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial will compare a typical 7-session therapeutic song-writing program with a waitlist-control group.
  Intervention group. The therapeutic song-writing program consists 7 session. One session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a helping professional who is familiar with music therapy will be recruited to run the therapeutic song-writing program at a collaborative social service centre and school. A standardized program manual is designed by the research team. The social workers and helping professionals who run the therapeutic song-writing program will receive training and supervision on conducting the therapeutic song-writing program by the research team.
Who Masked: Investigator
Masking Description: A research staff, who is blinded to the group allocation and does not involve in the delivery of group interventions, conduct the intervention outcomes assessment of the participants before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Therapeutic song-writing program
  Interventions: Behavioral: therapeutic song-writing program
- Waitlist Control Group (Other): Waitlist control group will receive will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive the same therapeutic song-writing program at a later stage.
  Interventions: Behavioral: Waitlist control group

INTERVENTIONS:
Behavioral: therapeutic song-writing program — The therapeutic song-writing program consists 7 session. One session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a helping professional who is familiar with music therapy will be recruited to run the therapeutic song-writing program at a collaborative social service centre and school. A standardized program manual is designed by the research team. The social workers and helping professionals who run the therapeutic song-writing program will receive training and supervision on conducting the therapeutic song-writing program by the research team.
  Arms: Intervention group
Behavioral: Waitlist control group — Waitlist control group will receive will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive the same therapeutic song-writing program at a later stage
  Arms: Waitlist Control Group

SUMMARY:
The research aims to investigate the effectiveness of the therapeutic song-writing program on young people with depressive symptoms.

This study adopts a multicentre randomized control trial two arms research design. A randomised controlled trial will compare a typical 7-session therapeutic song-writing program with a waitlist-control group to determine whether the 7-session therapeutic song-writing program can produce better outcomes for young people with depressive symptoms, including improvement in depressive symptoms, self-stigma, self-esteem, sense of hope and social support at post-intervention. The 7-session therapeutic song-writing program will be delivered by trained and experienced social workers and helping professionals who are familiar with music therapy. A research staff, who does not involve in the group allocation and delivery of group intervention, conduct the intervention outcomes assessment of the participants before and after the intervention. Standardized assessment tools are used to assess the intervention outcomes. The ethical considerations of this study were reviewed and approved by the Human and Artefacts Ethics Sub-Committee of the City University of Hong Kong in 2025.

DETAILED DESCRIPTION:
Mental health problems are very common among adolescents and youth in Hong Kong and worldwide. In Hong Kong, 24.4% of children and adolescents had at least one mental health problem in 2022. Mental health problems have negative effects on adolescents' health and academic performance, including suicide, alcohol and drug abuse, smoking, binge eating, diabetes, asthma and poor school performance. In particular, the risk of suicide among secondary school students is alarming in Hong Kong. 8.4%, 3.8% and 2.3% of secondary school students had a suicidal idea, plan or attempt in 2022, and the number of students who took their own lives in 2023 has increased by about 30% compared to the average of the past three years.

Psychosocial interventions have been shown to be effective in improving the mental health of adolescents and youth. Among the different types of psychosocial interventions, therapeutic song-writing has been shown to be effective in improving depressive symptoms and social support. Therapeutic song-writing facilitates ongoing self-exploration by enabling participants to explore, question, and challenge their sense of self, personal narratives, and ways of being. Meaning-making occurs in the outcomes and process of song-writing.

The therapeutic song-writing program, named Sound Bite, is a part of the "Everyone is a Hope Builder" organized by The Salvation Army of Hong Kong. As far as we know, no research study has been conducted on the effectiveness of a therapeutic song-writing program on improving the mental health of adolescents and youth in Hong Kong. Given this research gap, this research aims to explore the effectiveness of the therapeutic song-writing on young people with depressive symptoms.

Research Method This research study adopts mixed methods research design, involving both quantitative and qualitative study. The quantitative study aims to investigate the effectiveness of the therapeutic song-writing program for adolescent and youth people with depressive symptoms. The qualitative study aims to examine the benefits, advantages and limitations of the therapeutic song-writing program from the users' perspective. The ethical considerations of this study were reviewed and approved by the Human and Artefacts Ethics Sub-Committee of the City University of Hong Kong in 2025.

Quantitative Research Method Objective. This quantitative study aims to investigate the effectiveness of the therapeutic song-writing program for adolescents and youth with depressive symptoms.

Research Design. This study is a multicentre randomised waitlist-control study. Eligible participants will be recruited from local secondary schools and Salvation Army social service centres, through open recruitment via promotional activities and referrals from these units. A total of 120 participants will be recruited over a study period of approximately 18 months. Using block randomisation, 120 eligible participants will be randomly allocated in a 1:1 ratio to an intervention group or a waitlist control group. 60 participants in the intervention group will receive a therapeutic song-writing program. 60 participants on the waitlist-control group will not receive an intervention in the initial phase, but will receive the same therapeutic song-writing program at a later stage. 5 intervention groups and 5 waitlist-control groups will be conducted, with each intervention group consisting of 12 participants. A research assistant, blinded to randomised allocation, will conduct pre- and post-intervention outcome assessment using standardised assessment tools.

Hypotheses: After completing the therapeutic song-writing program, participants will show significantly greater improvement in depressive symptoms, self-stigma, self-esteem, sense of hope and social support at post-intervention.

Subject inclusion criteria:

1. aged between 13 to 24 years;
2. having mild to moderate depression and/or anxiety as assessed using a standardized assessment tool, i.e. Chinese Depression Anxiety Stress Scale-Youth (DASS-Y) with a DASS-Y Depression score between 5 and 12;
3. service users of The Salvation Army social service unit; and
4. giving informed consent to this research work. For those aged below 18, parental consent will be obtained.

Subject exclusion Criteria:

Those with severe depression (i.e. a DASS-Y Depression score ≥ 13) and severe anxiety (i.e. a DASS-Y Anxiety score ≥ 8) are excluded from this study.

Sample Size Estimation. The sample size of this study is estimated by using power analysis G*Power 3.1. Studies on interventions suggest a small to medium effect size on reducing depressive symptoms (Cohen's d ranges from 0.4 to 0.7). This study aims to demonstrate a medium effect size (i.e., Cohen's d = 0.5) with a statistical power of 0.80 for all intervention outcomes. A minimum sample size of 82 participants is required. Since a dropout rate of 30% is considered, a total of 120 participants are recruited.

Intervention group. The therapeutic song-writing program consists 7 session. One session will be conducted per week, with each session lasting for about 90 minutes. A social worker and a helping professional who is familiar with music therapy will be recruited to run the therapeutic song-writing program at a collaborative social service centre and school. A standardized program manual is designed by the research team. The social worker and a counsellor who run the therapeutic song-writing program will receive training and supervision on conducting the therapeutic song-writing program by the research team.

Waitlist-control group. Waitlist control group will receive will receive treatment as usual provided by the elderly centre, including recreational activities and interest classes, at the initial stage and will receive the same therapeutic song-writing program at a later stage.

Outcome assessment tools. The primary outcome is the reduction of depressive symptoms which is assessed by a 21-item Chinese Depression Anxiety Stress Scale-Youth (DASS-Y).

The secondary outcomes include improvement in self-stigma, self-esteem, hope and social support which are assessed by the following scales:

The Chinese Internalised Stigma of Mental Illness (ISMI) is a 10 -item self-reported scale to measure changes in self-stigma The Chinese Rosenberg Self-Esteem Scale (RSES) is a 10-item scale to assess participants' self-reported self-esteem The Chinese Hope Scale (HOPE) is a 12-item scale to assess participants' self-reported hope The Chinese Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item scale to assess participants' self-reported social support

Data analysis. An analysis will be performed in accordance with the intent-to-treat principle using multiple imputation method analysis for any missing data. For all analyses, two-tailed p values of < 0.05 is considered statistically significant. Data analyses will be performed using SPSS 29.0. Within group intervention effects are investigated using pair-sample t-test. Between group intervention effects are investigated using 2 (group) x 2 (time) repeated measures of one-way analysis of variance (ANOVA). Within and between group effect sizes are computed using Cohen's d, with values of 0.2, 0.5, and 0.8 considered as small, medium, and large respectively.

Fidelity of intervention. Standardized program manual of the therapeutic song-writing program will be developed by a project team of The Salvation Army. The program manuals will be reviewed by experts in song-writing programs. The social workers delivering the therapeutic song-writing program in this project will receive the program manuals, training and supervision from the project team to ensure that the intervention groups follow the program manual.

Qualitative Research Method Objective. This qualitative study aims to explore the benefits, advantages and limitations of the therapeutic song-writing program from the users' perspective.

Research Design. In the qualitative study, focus groups with purposive sampling will be conducted. Participants completing therapeutic song-writing programs will be selected to attend a focus group. Each focus groups will be facilitated by a research staff with an interview protocol developed for this study.

Data Collection. Participants will be asked questions such as the following: "In what ways, if any, did the intervention group help you to improve your mental health such as depression and anxiety"; "In what ways, if any, did the intervention group help you to improve self-esteem and build up a sense of hope?"; "What are the advantages and limitations, if any, of the intervention group?"; "and "Any suggestions, if any, for improving the intervention group?". The content of focus groups will be audio-recorded and transcribed into verbatim by the research team.

Data analysis. All transcripts of the focus groups will be imported and coded for data analysis. Reflective thematic analysis will be used to identify, analyse and report themes so that themes can be developed both inductively (i.e. data-driven) and deductively (i.e. theory-driven). The research team will systematically read and re-read the transcripts, following the six stages of analysis, including: (1) becoming familiar with the data, (2) generating codes, (3) constructing themes, (4) reviewing potential themes, (5) defining and naming themes, and (6) producing the report. Two research staff compare, review and refine the codes, categories and themes until they reach agreement.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 13 to 24 years;
2. having mild to moderate depression and/or anxiety as assessed using a standardized assessment tool, i.e. Chinese Depression Anxiety Stress Scale-Youth (DASS-Y) with a DASS-Y Depression score between 5 and 12;
3. service users of The Salvation Army social service unit; and
4. giving informed consent to this research work. For those aged below 18, parental consent will be obtained.

Exclusion Criteria:

Those with severe depression (i.e. a DASS-Y Depression score ≥ 13) and/or severe anxiety (i.e. a DASS-Y Anxiety score ≥ 8) are excluded from this study.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
The Chinese Depression Anxiety Stress Scale-Youth (DASS-Y) | It will be used before and after the intervention (over 7-weeks)
  The Chinese Depression Anxiety Stress Scale- Youth (DASS-Y; Cao et al., 2023) DASS-Y is a 21-item scale to assesses participants' self-reported depression, anxiety, and stress with good validity and reliability (Cronbach's α = 0.80 for the DASS-Y Anxiety subscale, 0.83 for the DASS-Y Depression subscale, 0.82 for the DASS Stress subscale, and 0.92 for the DASS-Y total scale). Each item (e.g. I felt down-hearted and blue) is scored from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The scores are summed over the items with higher scores indicating a higher severity of symptoms

SECONDARY OUTCOMES:
The Chinese Internalised Stigma of Mental Illness (ISMI) | It will be used before and after the intervention (over 7-weeks)
  The Chinese Internalized Stigma of Mental Illness (ISMI; Young et al., 2017) is a 10 -item self-reported scale to measure changes in self-stigma in four dimensions, i.e. shame/alienation (ISMI-SH), stereotype endorsement (ISMI-SE), perceived discrimination (ISMI-PD) and social withdrawal (IMIS-SW), with good validity and reliability (Cronbach's α = 0.93; 0.85; 0.75; 0.84 and for ISMI total scale, ISMI-SH, ISMI-SE, ISMI-PD, ISMI-SW). Each item (e.g. People discriminate against me because I have a mental illness) is rated with a score on a 4-point scale which ranges from "1" (strongly agree) to "4" (strongly disagree). Scores are averaged over the items, with higher scores indicating greater self-stigma.
Chinese Rosenberg Self-Esteem Scale (RSES) | It will be used before and after the intervention (over 7-weeks)
  The Chinese Rosenberg Self-Esteem Scale (RSES; Peng et al., 2024) is a 10-item scale to assess participants' self-reported self-esteem in two dimensions, i.e. self-worth (RSES-SW) and self-depreciation (RSES-SD) with good validity and reliability (Cronbach's α = 0.63; 0.74, and 0.81 for RSES, RESE-SW, and RSES-SD). Each item (e.g. I feel that I have a number of good qualities) is rated on a 4-point scale with scores ranging from "1" (strongly agree) to "4" (strongly disagree). The scores are summed over the items, with higher scores indicating better self-esteem.
Chinese Hope Scale (HOPE) | It will be used before and after the intervention (over 7-weeks)
  The Chinese Hope Scale (HOPE; Ho et al., 2012) is a 12-item scale to assess participants' self-reported hope in two dimensions, i.e., agency (i.e., goal-directed energy) and pathways (i.e., planning to accomplish goals) with good validity and reliability (Cronbach's α = 0.81; 0.70 and 0.76 for the Hope total scale, agency subscale and pathway subscale). Each item (e.g. I can think of many ways to get out of a jam) is answered using an 8-point scale ranging from "1" (definitely false) to "4" (definitely true). The scores are summed over the items, so that higher scores indicate a higher level of hope.
Chinese Multidimensional Scale of Perceived Social Support (MSPSS) | It will be used before and after the intervention (over 7-weeks)
  The Chinese Multidimensional Scale of Perceived Social Support (MSPSS; Yang et al., 2024) is a 12-item scale to assess participants' self-reported hope in three dimensions, i.e., family, friends, and significant others with good validity and reliability (Cronbach's α = 0.91, 0.77, 0.88, and 0.88 for the MSPSS total scale, family, friends, and significant others subscale). Each item (e.g. There is a special person with whom I can share joys and sorrows) is answered using a 7-point scale ranging from "1" (strongly disagree) to "7" (strongly agree). The scores are summed over the items, so that higher scores indicate greater social support

CONTACTS AND LOCATIONS:
Locations (1):
- City University of Hong Kong, Kowloon Tong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peng W, Zhou Y, Chu J, Liu Z, Zheng K, Yao S, Yi J. Factorial and Criterion Validities of the Chinese Version of Rosenberg Self-Esteem Scale Among Undergraduate Students. Psychol Res Behav Manag. 2024 Dec 5;17:4135-4144. doi: 10.2147/PRBM.S494452. eCollection 2024. PMID 39654814
- [Background] Cao CH, Liao XL, Gamble JH, Li LL, Jiang XY, Li XD, Griffiths MD, Chen IH, Lin CY. Evaluating the psychometric properties of the Chinese Depression Anxiety Stress Scale for Youth (DASS-Y) and DASS-21. Child Adolesc Psychiatry Ment Health. 2023 Sep 7;17(1):106. doi: 10.1186/s13034-023-00655-2. PMID 37679819
- [Background] Wang K, Shi HS, Geng FL, Zou LQ, Tan SP, Wang Y, Neumann DL, Shum DH, Chan RC. Cross-cultural validation of the Depression Anxiety Stress Scale-21 in China. Psychol Assess. 2016 May;28(5):e88-e100. doi: 10.1037/pas0000207. Epub 2015 Nov 30. PMID 26619091
- [Background] Li XH, Wong YI, Wu Q, Ran MS, Zhang TM. Chinese College Students' Stigmatization towards People with Mental Illness: Familiarity, Perceived Dangerousness, Fear, and Social Distance. Healthcare (Basel). 2024 Aug 27;12(17):1715. doi: 10.3390/healthcare12171715. PMID 39273739
- [Background] Ho SM, Ho JW, Bonanno GA, Chu AT, Chan EM. Hopefulness predicts resilience after hereditary colorectal cancer genetic testing: a prospective outcome trajectories study. BMC Cancer. 2010 Jun 11;10:279. doi: 10.1186/1471-2407-10-279. PMID 20537192
- [Background] Gee KA, Hawes V, Cox NA. Blue Notes: Using Songwriting to Improve Student Mental Health and Wellbeing. A Pilot Randomised Controlled Trial. Front Psychol. 2019 Mar 5;10:423. doi: 10.3389/fpsyg.2019.00423. eCollection 2019. PMID 30890979
- [Background] Duagi D, Carter B, Farrelly M, Lisk S, Shearer J, Byford S, James K, Brown JSL. Long-term effects of psychosocial interventions for adolescents on depression and anxiety: a systematic review and meta-analysis. EClinicalMedicine. 2024 Jan 5;68:102382. doi: 10.1016/j.eclinm.2023.102382. eCollection 2024 Feb. PMID 38273890
- [Background] Baker FA, Tamplin J, MacDonald RA, Ponsford J, Roddy C, Lee C, Rickard N. Exploring the Self through Songwriting: An Analysis of Songs Composed by People with Acquired Neurodisability in an Inpatient Rehabilitation Program. J Music Ther. 2017 Mar 1;54(1):35-54. doi: 10.1093/jmt/thw018. PMID 28391303